CLINICAL TRIAL: NCT01723410
Title: Neural and Physiological Responses to Real-World Experiences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Naomi Eisenberger, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GGSC-GRAT
Record Dates: First submitted 2012-11-01; First posted 2012-11-07 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Gene Expression
MeSH Terms: interventions — Artifacts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Writing condition (Experimental): Subjects will be asked to write about other individuals in their lives.
  Interventions: Behavioral: Writing about people
- Writing (Placebo Comparator): Subjects will be asked to write about places or objects in their lives.
  Interventions: Other: Writing about places, objects

INTERVENTIONS:
Behavioral: Writing about people — Subjects will be asked to write about other people in their lives once a week for 6-weeks.
  Arms: Writing condition
Other: Writing about places, objects
  Arms: Writing

SUMMARY:
UCLA researchers looking for healthy individuals (aged 35-50) who have a home computer with internet access, are not pregnant, planning to become pregnant, or currently breastfeeding (if female), to participate in a study investigating whether real-world experiences alter the brain and body. This study takes place over an eight week period and involves providing the names of 8 close friends or family members, completing a neuroimaging session, providing blood and saliva (for genetic analysis), and a 6-week period in which participants login twice a week to complete online questionnaires. Compensation is up to $210 for those who complete all aspects of the study. Please email realworld.ucla@gmail.com for more information.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 35-50

Exclusion Criteria:

Following a structured telephone interview, prospective participants with the following conditions will not be able to participate:

1. claustrophobia, left-handedness, or presence of metal in their body (for the neuroimaging procedures),
2. possible presence of a depressive disorder, which may interfere with the gratitude intervention (assessed by the Patient Health Questionnaire; Spitzer et al., 1999),
3. regular use of medications that may impact inflammatory processes (anti-inflammatory drugs, steroids, opioids),
4. current smokers or excessive caffeine users (> 600 mg/day) because of known effects on inflammation, and
5. pregnancy (which would affect oxytocin gene expression).

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
inflammatory gene expression | baseline, six weeks post manipulation
  Changes in inflammatory gene expression from pre- to post-intervention.

SECONDARY OUTCOMES:
neural activity | baseline, six weeks post-intervention
  Changes in neural activity from pre- to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi I Eisenberger, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA CTRC & Brain Mapping Center, Los Angeles, California, United States